CLINICAL TRIAL: NCT01218490
Title: Pelvic and Aortic-cava Lymphadenectomy Randomized Phase III for Advanced Ovarian Cancer
Brief Title: Pelvic and Aortic-cava Lymphadenectomy Randomized for Ovarian Cancer
Acronym: CARACO
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: qualitative analysis of the study database
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SC 07/12-H
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Ovarian Cancer
Keywords: surgery; ovarian cancer; lymphadectomy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lymphadenectomy (Experimental): after surgery of the ovarian cancer, patient will have Pelvis and aortic-cava lymphadenectomy
  Interventions: Procedure: ovarian cancer surgery
- no lymphadectomy (No Intervention): after surgery, the patient will not have pelvic and aortic-cave lymphadenectomy

INTERVENTIONS:
Procedure: ovarian cancer surgery
  Arms: lymphadenectomy

SUMMARY:
It is a multicenter randomized trial of superior cleaning compared the absence of dissection in stage III patients with optimal surgical resection without retroperitoneal lymph node palpable.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Karnofsky> 80, or ASA I-II
* Primary ovarian adenocarcinoma, or primitive peritoneal
* No retroperitoneal lymph node> 2cm (CT; MRI)
* Complete surgical staging
* Stage III-IV FIGO classification
* Indication of systemic chemotherapy before surgery or post surgery

Exclusion Criteria:

* Non Invasive Cancer
* non-epithelial or borderline cancer
* Pregnancy
* Previous pelvic lymphadenectomy or aortic-cava for a disease other than ovarian cancer
* Contraindication to Platinum and Paclitaxel
* Borderline Ovarian Tumor
* tumor recurrence
* Incomplete surgery, resectable lesion, Surgery sub optimal (R> 1cm)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2008-12-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
survival with out recurrence | 5 years

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - Clinique Sainte Thérèse, Amiens
  - Centre Paul Papin, Angers
  - Hospital, Angers
  - Hospital, Brest
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre G F Leclerc, Dijon
  - Hospital, Lyon
  - Institut Paoli Calmette, Marseille
  - Centre Val d'Aurelle, Montpellier
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital des Diaconesses, Paris
  - Clinique Mutualiste, Rennes
  - Hopital, Rennes
  - Centre René Huguenin, Saint-Cloud
  - Institut Cancerologie de l'Ouest, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Hôpital Bretonneau, Tours